CLINICAL TRIAL: NCT04908683
Title: A Randomized, Double-blind, Placebo-controlled Phase 3 Efficacy Study of an Ad26.RSV.preF-based Vaccine in the Prevention of Lower Respiratory Tract Disease Caused by RSV in Adults Aged 60 Years and Older
Brief Title: A Study of an Adenovirus Serotype 26 Pre-fusion Conformation-stabilized F Protein (Ad26. RSV. preF) Based Respiratory Syncytial Virus (RSV) Vaccine in the Prevention of Lower Respiratory Tract Disease in Adults Aged 60 Years and Older
Acronym: EVERGREEN
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR108959; 2020-005458-97 (EudraCT Number); VAC18193RSV3001 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Results first posted 2024-02-08 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Respiratory Syncytial Viruses; Lower Respiratory Tract Disease
Keywords: Acute Respiratory Infections; Vaccine; Ad26.RSV.preF-based Vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Respiratory Syncytial Virus (RSV) vaccine (Experimental): All participants in the active group will receive a single dose intramuscular (IM) injection of study vaccine on Day 1.
  Interventions: Biological: Adenovirus serotype 26 (Ad26)-based respiratory syncytial virus (RSV). preF
- Group 2: Placebo (Placebo Comparator): All participants in the placebo group will receive a single IM injection of matching placebo on Day 1.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Adenovirus serotype 26 (Ad26)-based respiratory syncytial virus (RSV). preF — Participants will receive a single IM injection of an RSV vaccine.
  Arms: Group 1: Respiratory Syncytial Virus (RSV) vaccine
Biological: Placebo — Participants will receive a single IM injection of matching placebo.
  Arms: Group 2: Placebo

SUMMARY:
The study will enroll up to 27,200 participants in order to demonstrate the efficacy of the active Ad26.RSV.preF-based study vaccine in the prevention of Reverse Transcription Polymerase Chain Reaction (RT-PCR) confirmed Respiratory Syncytial Virus (RSV)-mediated Lower Respiratory Tract Disease (LRTD) when compared to placebo in adults aged 60 years and above.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to work with smartphones/tablets/computers
* From the time of vaccination through 3 months after vaccination, participant agrees not to donate blood
* Must be willing to provide verifiable identification, has means to be contacted and to contact the investigator during the study
* Before randomization, a participant must be: a. postmenopausal (postmenopausal state is defined as no menses for 12 months without an alternative medical cause); and b. not intending to conceive by any methods
* Participants must sign an Inform Consent Form (ICF) indicating that the participant understands the purpose, procedures and potential risks and benefits of the study, and is willing to participate in the study

Exclusion Criteria:

* Has a serious clinically unstable condition, (example, end-stage renal disease with or without dialysis, clinically unstable cardiac disease), Alzheimer's disease, or any other condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (example, compromise well-being) or that could prevent, confound, or limit the protocol specified assessments
* History of malignancy within 5 years before screening not in the following categories: a. Participants with squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix may be enrolled at the discretion of the investigator; b. Participants with a history of malignancy within 5 years, which is considered cured with minimal risk of recurrence per investigator's judgement, can be enrolled
* Had major surgery (example, major cardiopulmonary or abdominal operations) as per the investigator's judgment within 4 weeks before vaccination, or will not have fully recovered from surgery, or has major surgery planned during the time the participant is expected to participate in the study
* Employee of the investigator or study site, with direct involvement in the proposed study or other studies under the direction of that investigator or study site, as well as family members of the employees or the investigator, or an employee of the sponsor
* Contraindication to Intramuscular (IM) injections and blood draws (example, bleeding disorders)
* Known or suspected allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine components (including any of the constituents of the study vaccine)

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25236 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (272):
- United States (156):
  - Central Research Associates, Inc., Birmingham, Alabama
  - Synexus Clinical Research US Inc, Birmingham, Alabama
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Optimal Research, Huntsville, Alabama
  - Coastal Clinical Research, Inc, Mobile, Alabama
  - Synexus Clinical Research US Inc, Chandler, Arizona
  - Hope Research Institute, Peoria, Arizona
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Medpharmics, LLC, Phoenix, Arizona
  - Clinical Research Consortium Arizona, Tempe, Arizona
  - Synexus Clinical Research US Inc, Tucson, Arizona
  - Baptist Health Center For Clinical Research, Little Rock, Arkansas
  - Rancho Paseo Medical Group, Banning, California
  - Hope clinical Research LLC, Canoga Park, California
  - Synexus Clinical Research US Inc, Cerritos, California
  - eStudySite, Chula Vista, California
  - Velocity Clinical Research, San Diego, La Mesa, California
  - Paradigm Clinical Research Centers, Inc., Redding, California
  - Optimal Research, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Synexus Clinical Research US Inc, Vista, California
  - Synexus Clinical Research US Inc, Aurora, Colorado
  - Tekton Research Inc., Fort Collins, Colorado
  - Tekton Research Inc., Longmont, Colorado
  - Paradigm Clinical Research Centers, Inc., Wheat Ridge, Colorado
  - JEM Research LLC, Atlantis, Florida
  - Clinical Research of South Florida, an AMR Company, Coral Gables, Florida
  - Prestige Clinical Research Center, Inc., Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Velocity Clinical Research, Inc., Edgewater, Florida
  - AMR Fort Myers Clinical Physiology Associates, an AMR company, Fort Myers, Florida
  - Velocity Clinical Research, Hallandale Beach, Hallandale, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Altus Research, Inc, Lake Worth, Florida
  - Accel Research Sites, Lakeland, Florida
  - Compass Research LLC, Leesburg, Florida
  - Optimal Research, Melbourne, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Suncoast Research Associates, LLC, Miami, Florida
  - Clinical Site Partners, LLC, Miami, Florida
  - Healthcare Clinical Data Inc., North Miami, Florida
  - Harmony Clinical Research Inc, North Miami Beach, Florida
  - Clinical NeuroScience Solutions Inc, Orlando, Florida
  - Headlands Research Orlando, Orlando, Florida
  - Synexus Clinical Research US Inc, Orlando, Florida
  - Synexus Clinical Research US Inc, Pinellas Park, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Sandhill Research, St. Petersburg, Florida
  - DBC Research, Tamarac, Florida
  - Palm Beach Research Center, West Palm Beach, Florida
  - Synexus Clinical Research US Inc, Atlanta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - Accel Research Sites, Eatonton, Georgia
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Advanced Clinical Research, Boise, Idaho
  - Christie Clinic, Champaign, Illinois
  - Synexus Clinical Research US Inc, Chicago, Illinois
  - Optimal Research, Peoria, Illinois
  - Medisphere Medical Research Center, Llc, Evansville, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - Buynak Clinical Research, Valparaiso, Indiana
  - The Iowa Clinic, P.C., West Des Moines, Iowa
  - Heartland Research Associates, LLC, Augusta, Kansas
  - Johnson County Clin-Trials, Lenexa, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Clinical Research, Wichita, Kansas
  - Central Kentucky Research Associates, Inc., Lexington, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Medpharmics, LLC, Kenner, Louisiana
  - Medpharmics, LLC, Lafayette, Louisiana
  - Centex Studies, Inc., Lake Charles, Louisiana
  - Clinical Trials of America, Monroe, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - AMR New Orleans, Formerly New Orleans Center for Clinical Research - New Orleans, an AMR company, New Orleans, Louisiana
  - Central Maine Medical Center, Lewiston, Maine
  - Centennial Medical Group, Elkridge, Maryland
  - Optimal Research, Rockville, Maryland
  - Synexus Clinical Research US Inc, Richfield, Minnesota
  - MedPharmics - Biloxi, Biloxi, Mississippi
  - Jefferson City Medical Group Family, Jefferson City, Missouri
  - The Center for Pharmaceutical Research (CPR), Kansas City, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Synexus Clinical Research US Inc, St Louis, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Meridian Clinical Research, LLC, Norfolk, Nebraska
  - Meridian Clinical Research - Omaha, Omaha, Nebraska
  - Synexus Clinical Research US Inc, Omaha, Nebraska
  - Synexus Clinical Research US Inc, Henderson, Nevada
  - Clinical Research Consortium, an AMR company, Las Vegas, Nevada
  - Medpharmics, LLC, Albuquerque, New Mexico
  - Meridian Clinical Research, LLC, Endwell, New York
  - Regional Clinical Research, Inc., Endwell, New York
  - Synexus Clinical Research US Inc, Manhattan, New York
  - Harlem Hospital Center, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - CHEAR Center, LLC, The Bronx, New York
  - Accellacare Research of Cary, Cary, North Carolina
  - American Health Network, LLC, Charlotte, North Carolina
  - M3-Emerging Medical Research, Durham, North Carolina
  - Medication Management LLC, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare Research of Cary, Raleigh, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Trial Management Associates, LLC, Wilmington, North Carolina
  - Accellacare Research of Cary, Winston-Salem, North Carolina
  - Synexus Clinical Research US Inc, Akron, Ohio
  - Synexus Clinical Research US Inc, Cincinnati, Ohio
  - Velocity Clinical Research, Cincinnati, Ohio
  - Rapid Medical Research, Cleveland, Ohio
  - Synexus Clinical Research US Inc, Columbus, Ohio
  - Lynn Institute of Norman, Norman, Oklahoma
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tekton Research Inc., Yukon, Oklahoma
  - Clinical Research Institute of Southern Oregon, P.C., Grants Pass, Oregon
  - Clinical Research Institute of Southern Oregon, P.C., Medford, Oregon
  - Preferred Primary Care Physicians Research, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians Research, Uniontown, Pennsylvania
  - Omega Medical Research, Warwick, Rhode Island
  - Synexus Clinical Research US Inc, Anderson, South Carolina
  - Velocity Clinical Research, Inc., Gaffney, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - PMG Research of Charleston, LLC, Mt. Pleasant, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - VitaLink Research Spartanburg, Spartanburg, South Carolina
  - Meridian Clinical Research - Dakota Dunes, Dakota Dunes, South Dakota
  - PMG Research of Bristol, Bristol, Tennessee
  - VGR & NOCCR - Knoxville, Knoxville, Tennessee
  - Clinical Research Associates Inc, Nashville, Tennessee
  - Central Texas Clinical Research, Austin, Texas
  - Optimal Research, Austin, Texas
  - Tekton Research Inc., Austin, Texas
  - Tekton Research Inc., Beaumont, Texas
  - Advanced Clinical Research, Cedar Park, Texas
  - Synexus Clinical Research US Inc, Dallas, Texas
  - North Texas Infectious Diseases Consultants, Dallas, Texas
  - Vilo Research Group Inc, Houston, Texas
  - Texas Center for Drug Development Inc, Houston, Texas
  - Research Your Health, Plano, Texas
  - Clinical Trials of Texas Inc, San Antonio, Texas
  - Synexus Clinical Research US Inc, San Antonio, Texas
  - Tekton Research Inc., San Antonio, Texas
  - DM Clinical Research, Tomball, Texas
  - Martine Diagnostic Clinic, Tomball, Texas
  - Synexus Clinical Research US Inc, Layton, Utah
  - Synexus Clinical Research US Inc, Murray, Utah
  - Advanced Clinical Research, West Jordan, Utah
  - Charlottesville Medical Research Center, LLC, Charlottesville, Virginia
  - Spectrum Medical, Inc, Danville, Virginia
  - Health Research of Hampton Roads, Inc, Newport News, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - Amherst Family Practice, PC, Winchester, Virginia
- Australia (4):
  - Paratus Clinical Canberra Clinic, Bruce
  - Northside Health, Coffs Harbour
  - Paratus Clinical Kanwal Clinic, Kanwal
  - Mater Hospital Brisbane, South Brisbane
- Brazil (5):
  - UFRR - Universidade Federal de Roraima, Boa Vista
  - CMIP - Centro Mineiro de Pesquisa Ltda, Juiz de Fora
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - CPQuali Pesquisa Clinica LTDA ME, São Paulo
- Canada (10):
  - Okanagan Clinical Trials, Kelowna, British Columbia
  - LMC Clinical Research dba Manna Research Inc. Burlington, Burlington, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - LMC Clinical Research dba Manna Research Inc. Toronto, Toronto, Ontario
  - LMC Clinical Research dba Manna Research Inc. Quebec City, Lévis, Quebec
  - LMC Clinical Research dba Manna Research Inc. Montreal, Pointe-Claire, Quebec
  - DIEX Recherche Quebec Inc., Québec, Quebec
  - DIEX Recherche Joliette Inc., Saint-Charles-Borromée, Quebec
  - DIEX Recherche Sherbrooke Inc, Sherbrooke, Quebec
  - DIEX Recherche Victoriaville Inc., Victoriaville, Quebec
- Chile (3):
  - CENRESIN, Quilota
  - Centro de Estudios Clínicos e Investigación Médica (CeCim), Santiago
  - Centro de Investigacion del Maule, Talca
- China (3):
  - Donghai County Center for Disease prevention and Control, Lianyungang
  - Funing County Center for Disease Control and Prevention, Yancheng
  - Binhai County Center for Disease Control and Prevention, Yancheng
- Estonia (3):
  - OU Innomedica, Tallinn
  - Center for Clinical and Basic Research, Tallinn
  - Clinical Research Centre, Tartu
- Finland (10):
  - Espoon rokotetutkimusklinikka, Espoo
  - Etelä-Helsingin rokotetutkimusklinikka, Helsinki
  - Itä-Helsingin rokotetutkimusklinikka, Helsinki
  - Järvenpään rokotetutkimusklinikka, Jarvenpaa
  - Kokkolan rokotetutkimusklinikka, Kokkola
  - Oulun rokotetutkimusklinikka, Oulu
  - Porin rokotetutkimusklinikka, Pori
  - Seinäjoen rokotetutkimusklinikka, Seinäjoki
  - Tampereen rokotetutkimusklinikka, Tampere
  - Turun rokotetutkimusklinikka, Turku
- New Zealand (13):
  - Southern Clinical Trials Totara Clinical Research, Auckland
  - Southern Clinical Trials, Waitemata, Auckland
  - Optimal Clinical Trials, Auckland
  - Southern Clinical Trials, Christchurch, Christchurch
  - Lakeland Clinical Trials, Hamilton
  - P3 Research Ltd, Havelock North
  - Southern Clinical Trials Tasman, Main Road Stoke
  - P3 Research Ltd, Palmerston North
  - P3 Research Limited Kapiti, Paraparaumu
  - Lakeland Clinical Trials, Rotorua
  - P3 Research Ltd, Tauranga
  - Lakeland Clinical Trials, Upper Hutt
  - P3 Reaearch Wellington, Wellington
- Poland (13):
  - Synexus Polska Sp. z o.o. Oddzial w Czestochowie, Częstochowa
  - Synexus Polska Sp. z o.o. Oddzial w Gdansku, Gdansk
  - Synexus Scm Sp Z o o Oddzial Gdynia, Gdynia
  - Synexus Polska Sp z o o Oddzial w Katowicach, Katowice
  - Synexus Polska Sp z o o, Lodz
  - KO MED Centra Kliniczne LUBLIN, Lublin
  - Synexus Polska Sp. z.o.o. Oddzial w Poznaniu, Poznan
  - KO MED Centra Kliniczne Pulawy, Puławy
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Synexus Polska Sp z o o Oddzial w Warszawie, Warsaw
  - Synexus Polska Sp z o o Oddzial we Wroclawiu, Wroclaw
  - KO MED Centra Kliniczne Zamosc, Zamość
- South Africa (23):
  - Iatros International, Bloemfontein
  - Josha Research, Bloemfontein
  - Madibeng Centre for Research, Brits
  - Synexus Helderberg Clinical Research Centre, Cape Town
  - TREAD Research Tygerberg Hospital, Cape Town
  - TASK Central, Cape Town
  - Tiervlei Trial Centre, Cape Town
  - Allergy Immunology Unit, Cape Town
  - Synergy Biomed Research Institute (SBRI), East London
  - TASK Central, George
  - CRISMO Bertha Gxowa Research Centre, Johannesburg
  - Worthwhile Clinical trials, Johannesburg
  - Clinresco Centres Pty Ltd, Johannesburg
  - DJW Research, Krugersdorp
  - Stanza Clinical Research Centre : Mamelodi, Mamelodi East
  - Newtown Clinical Research, Newtown
  - Paarl Research Centre, Paarl
  - Global Clin Trials Pretoria, Pretoria
  - Synexus Watermeyer, Pretoria
  - The Aurum Institute Rustenburg Clinical Research Site, Rustenburg
  - REIMED Vosloorus, Vosloorus
  - Welkom Clinical Trial Centre, Welkom
  - Be Part Yoluntu Centre, Western Cape
- Taiwan (8):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital- Linkou, Taoyuan
- Thailand (6):
  - Royal Thai Army, Afrims, Bangkok
  - The Vaccine Trial Center(VTC), Faculty of Tropical Medicine, Bangkok
  - Siriraj Hospital, Bangkok
  - Srinagarind Hospital, Khon Kaen
  - Maharaj Nakorn Chiang Mai hospital Faculty of Medicine, Muang
  - King Chulalongkorn Memorial Hospital, Pathumwan
- United Kingdom (15):
  - Synexus Midlands Clinical Research Centre, Birmingham
  - FutureMeds Soho Health Centre, Birmingham
  - Bradford Royal Infirmary, Bradford
  - FutureMeds Bridle Clinic, Bromborough
  - Synexus Wales Clinical Research Center, Cardiff
  - Synexus Lancashire Clinical Research Centre, Chorley
  - Panthera Biopartners, Glasgow
  - Synexus Scotland Clinical Research Centre, Glasgow
  - Synexus Hexham General Hospital, Hexham
  - Synexus Merseyside Clinical Research Centre, Liverpool
  - Synexus Manchester Clinical Research Center, Manchester
  - North Manchester General Hospital, Manchester
  - Panthera Biopartners, Preston
  - Panthera Biopartners, Reading
  - University Hospital of North Tees, Stockton-on-Tees

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Langer S, Holzapfel S, August L, Badura A, Wellmann S, Mack I. Parental knowledge and attitudes to infant immunization in the context of RSV: All about confidence? Vaccine. 2024 Oct 3;42(23):126050. doi: 10.1016/j.vaccine.2024.06.018. Epub 2024 Jun 19. PMID 38902186

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Ad26.RSV.preF and RSV preF Protein: Participants received a single intramuscular (IM) injection containing a mixture of adenovirus serotype 26 respiratory syncytial virus pre-fusion conformation stabilized F-protein (Ad26.RSV.preF) at a dose of 1*10^11 viral particles (vp) and RSV preF protein 150 micrograms (mcg) on Day 1.
- Group 2: Placebo: Participants received a single IM injection of matching placebo on Day 1.
Period: Overall Study
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Started | 16817 | 8419
Randomized and Vaccinated | 16709 | 8367
Completed | 124 | 59
Not Completed | 16693 | 8360
Not completed — Failure to meet continuation criteria | 34 | 22
Not completed — Initiated prohibited medication | 3 | 0
Not completed — Randomized by mistake | 1 | 0
Not completed — Lost to Follow-up | 679 | 341
Not completed — Participant met eligibility criteria but were not needed | 3 | 1
Not completed — Physician Decision | 44 | 35
Not completed — Technical problems | 12 | 9
Not completed — Withdrawal by legally authorized representative | 1 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 1188 | 570
Not completed — Site Closure by Sponsor | 6 | 3
Not completed — Adverse Event | 21 | 11
Not completed — Death | 101 | 61
Not completed — Sponsor's decision | 14398 | 7205
Not completed — Other | 92 | 50
Not completed — Randomized not vaccinated | 108 | 52

BASELINE CHARACTERISTICS:
Population: Baseline characteristics data were analyzed on full analysis set (FAS) which included all participants with a documented vaccine administration, regardless of the occurrence of protocol deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo | Total
Number analyzed (Participants) | 16709 | 8367 | 25076
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (5.24) | 70.2 (5.23) | 70.2 (5.24)
Age, Customized [Count of Participants; unit: Participants]
  Adults (60-64 years) | 1472 | 740 | 2212
  From 65 to 84 years | 15053 | 7534 | 22587
  85 years and over | 184 | 93 | 277
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 9063 | 4452 | 13515
  Male | 7645 | 3913 | 11558
  Others | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1555 | 741 | 2296
  Not Hispanic or Latino | 14903 | 7496 | 22399
  Unknown or Not Reported | 251 | 130 | 381
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 58 | 17 | 75
  Asian | 1757 | 897 | 2654
  Native Hawaiian or Other Pacific Islander | 98 | 49 | 147
  Black or African American | 1820 | 935 | 2755
  White | 12649 | 6297 | 18946
  More than one race | 189 | 101 | 290
  Unknown or Not Reported | 138 | 71 | 209

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of Reverse Transcriptase Polymerase Chain Reaction (RT-PCR)-Confirmed Respiratory Syncytial Virus (RSV) Mediated Lower Respiratory Tract Disease (LRTD)
Description: Number of participants with first occurrence of RT-PCR-confirmed RSV mediated LRTD according to protocol defined criteria were reported. A participant was considered to have RT-PCR-confirmed RSV-mediated LRTD if the following criteria were met: new onset or worsening from baseline of 3 or more of the symptoms as captured on the respiratory infection intensity and impact questionnaire (RiiQ, version 2) at the same assessment time point: cough, short of breath, coughing up phlegm (sputum), and wheezing and confirmation of RSV by RT-PCR in one or more of the nasal swabs, or in the sputum sample. RiiQ symptom scale was a 13-item questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The total LRTD symptom score was calculated as the mean of the 4 lower respiratory scores (cough, short of breath, coughing up phlegm [sputum] and wheezing).
Time Frame: From Baseline (Day 1) up to 12 months
Population: Per-protocol efficacy (PPE) population included all randomized and vaccinated participants, excluding those with major protocol deviations (MPDs) expecting to impact the efficacy outcomes. Participants with an RSV onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 16263 | 8152
Participants | 44 | 63

2. Secondary Outcome: Number of Participants With First Occurrence of Any RT-PCR-Confirmed RSV-mediated Acute Respiratory Infection (ARI)
Description: A participant was considered to have RT-PCR-confirmed RSV-mediated ARI if the following protocol defined criteria were met: ARI episode initiated by the participant and confirmed by the site with symptoms consistent with an ARI (new symptoms or worsening from baseline of at least one of the symptoms as captured on the RiiQ): sore throat, nasal congestion, cough, short of breath, coughing up phlegm (sputum), wheezing and confirmation of RSV by RT-PCR in one or more of the nasal swabs, or in the sputum sample. RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The total ARI symptom score was calculated as the mean of the 4 lower respiratory scores (cough, short of breath, coughing up phlegm [sputum] and wheezing).
Time Frame: From Baseline (Day 1) up to 12 months
Population: PPE population included all randomized and vaccinated participants, excluding those with MPDs expecting to impact the efficacy outcomes. Participants with an RSV onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 16263 | 8152
Participants | 77 | 101

3. Secondary Outcome: Number of Participants With First Occurrence of RT-PCR-Confirmed RSV Mediated LRTD During the Second Year
Description: Number of participants with first occurrence of any RT-PCR-confirmed RSV mediated LRTD during the second year were reported. A participant was considered to have RT-PCR-confirmed RSV-mediated LRTD if the following criteria were met: new onset or worsening from baseline of 3 or more of the symptoms as captured on the RiiQ, version 2 at the same assessment time point: cough, short of breath, coughing up phlegm (sputum), and wheezing and confirmation of RSV by RT-PCR in one or more of the nasal swabs, or in the sputum sample. RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The total LRTD symptom score was calculated as the mean of the 4 lower respiratory scores (cough, short of breath, coughing up phlegm [sputum] and wheezing).
Time Frame: From Month 12 up to Month 24
Population: PPE population included all randomized and vaccinated participants, excluding those with MPDs expecting to impact the efficacy outcomes. Participants with an RSV onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 10031 | 5011
Participants | 16 | 29

4. Secondary Outcome: Number of Participants With First Occurrence of Any RT-PCR-Confirmed RSV Mediated ARI During the Second Year
Description: A participant was considered to have RT-PCR-confirmed RSV-mediated ARI according to protocol defined criteria were reported. A participant was considered to have RT-PCR-confirmed RSV-mediated ARI if the following criteria were met: ARI episode initiated by the participant and confirmed by the site with symptoms consistent with an ARI (new symptoms or worsening from baseline of at least one of the symptoms as captured on the RiiQ): sore throat, nasal congestion, cough, short of breath, coughing up phlegm (sputum), wheezing and confirmation of RSV by RT-PCR in one or more of the nasal swabs, or in the sputum sample. RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. The total ARI symptom score was calculated as the mean of the 4 lower respiratory scores (cough, short of breath, coughing up phlegm [sputum] and wheezing).
Time Frame: From Month 12 up to Month 24
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 10031 | 5011
Participants | 39 | 44

5. Secondary Outcome: Number of Participants With First Occurrence of Predefined Clinically Relevant Disease Associated With RT-PCR-Confirmed RSV-Mediated ARI Over the Whole Study
Description: A participant was considered to have clinically relevant disease with specific parameters associated with an RT-PCR-confirmed RSV-mediated ARI if the following criteria were met: the participant had an RT-PCR-confirmed RSV-mediated ARI: ARI episode initiated by the participant and confirmed by the site with symptoms consistent with an ARI (new symptoms or worsening from baseline of at least one of the symptoms as captured on the RiiQ): sore throat, nasal congestion, cough, short of breath, coughing up phlegm (sputum), wheezing and confirmation of RSV by RT-PCR in one or more of the nasal swabs, or in the sputum sample; any of the following associated with ARI: hospitalization, emergency department visit, per clinical judgement of complications, decreased oxygen saturation, tachypnea, need of supplemental oxygen, hypotension, pulmonary function test and arterial blood gas result.
Time Frame: Baseline (Day 1) up to 24 months
Population: PPE population is defined as population included all randomized and vaccinated participants, excluding those with MPDs expecting to impact the efficacy outcomes. Participants with an RSV onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 16263 | 8152
Participants | 4 | 11

6. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: Number of participants with SAEs were reported. An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a pharmaceutical (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. An SAE is any untoward medical occurrence that at any dose may result in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a suspected transmission of any infectious agent via a medicinal product.
Time Frame: 28 days post vaccination on Day 1 (Day 29); First year follow-up (from Day 29 up to 6 months, that is, up to Day 154)
Population: Full analysis set (FAS) included all participants with a documented vaccine administration, regardless of the occurrence of protocol deviations. Here, 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 16709 | 8367
Participants
  28 days post vaccination on Day 1 | 119 | 53
  First year follow-up: number analyzed (Participants) | 16532 | 8275
  First year follow-up | 446 | 239

7. Secondary Outcome: Number of Participants With Potential Adverse Events of Special Interest (AESIs)
Description: Number of participants with potential AESIs were reported. AESIs were significant AEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. AESIs were embolic and thrombotic events, hematopoietic thrombocytopenia, and cerebral hemorrhage.
Time Frame: 28 days post vaccination on Day 1 (Day 29); First year follow-up (from Day 29 up to 6 months, that is, up to Day 154)
Population: FAS included all participants with a documented vaccine administration, regardless of the occurrence of protocol deviations. Here, 'n' (number analyzed) represents number of participants who were evaluable for specified timepoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 16709 | 8367
Participants
  28 days post vaccination on Day 1 | 25 | 4
  First year follow-up: number analyzed (Participants) | 16532 | 8275
  First year follow-up | 71 | 35

8. Secondary Outcome: Number of Participants With Solicited Local Adverse Events (AEs) up to 7 Days After Vaccination
Description: Number of participants with solicited local AEs 7 days post vaccination were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited local AEs were precisely defined events that participants were specifically asked about and which were noted by participants in the diary. Solicited local AEs included erythema, swelling, and pain/tenderness at the study vaccine injection site, were used to assess the reactogenicity of the study vaccine and were pre-defined local (injection site). All solicited AEs at the injection site (local) were considered related to the study vaccine administration.
Time Frame: Up to Day 7 post vaccination on Day 1 (up to Day 8)
Population: The safety subset included all participants that consented to the collection of AEs (solicited AEs for up to 7 days after vaccination). Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 2305 | 1155
Participants | 1076 | 169

9. Secondary Outcome: Number of Participants With Solicited Systemic AEs up to 7 Days After Vaccination
Description: Number of participants with solicited systemic AEs 7 days post vaccination were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Solicited systemic AEs included fatigue, headache, myalgia, nausea, pyrexia, for which participants were specifically questioned and which were noted by participants in their participant diary for 7 days post vaccination (day of vaccination and the subsequent 7 days).
Time Frame: Up to Day 7 post vaccination on Day 1 (up to Day 8)
Population: The safety subset (a subset of FAS) included all participants that consented to the collection of AEs (solicited AEs for up to 7 days after vaccination). Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 2305 | 1155
Participants | 1018 | 236

10. Secondary Outcome: Number of Participants With Unsolicited AEs up to 28 Days After Vaccination
Description: Number of participants with unsolicited AEs 28 days post vaccination were reported. An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. Unsolicited adverse events included all adverse events for which the participant was not specifically questioned in the subject diary.
Time Frame: Up to 28 days post vaccination on Day 1 (up to Day 29)
Population: The safety subset (a subset of FAS) included all participants that consented to the collection of AEs (unsolicited AEs for 28 days after vaccination). Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 2330 | 1165
Participants | 554 | 206

11. Secondary Outcome: Respiratory Syncytial Virus (RSV) A2 Strain Neutralization Antibody Titers at 14 Days Post Vaccination
Description: RSV A2 strain neutralizing antibody titers of the vaccine-induced immune response was assessed through virus neutralization assay.
Time Frame: At 14 Days post vaccination on Day 1 (Day 15)
Population: Per-protocol Immunogenicity (PPI) population included all randomized and vaccinated participants who were part of the immunogenicity subset (consisted of at least 360 participants, of whom ~50% were at increased risk for severe RSV disease and ~50% were 75 years or older) and for whom immunogenicity data were available. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 219 | 108
Titers | 7194 [6394 to 8093] | 537 [455 to 634]

12. Secondary Outcome: Geometric Mean Titers (GMTs) of Prefusion F-protein (Pre-F) Antibodies Immunoglobulin G (IgG) as Assessed by Enzyme-linked Immunosorbent Assay (ELISA) at 14 Days Post Vaccination
Description: GMTs of preF antibodies IgG at 14 days after the administration of Ad26.RSV.preF-based vaccine as assessed by ELISA were reported.
Time Frame: At 14 days post vaccination on Day 1 (Day 15)
Population: PPI population included all randomized and vaccinated participants who were part of the immunogenicity subset and for whom immunogenicity data were available. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 219 | 108
Titers | 4932 [4477 to 5433] | 410 [348 to 484]

13. Secondary Outcome: T-cell Interferon (IFN) Gamma Responses to Respiratory Syncytial Virus (RSV) F Protein Peptides Analyzed by Enzyme-linked Immunospot Assay (ELISpot)
Description: T-cell IFN gamma responses to RSV F protein specific peptides at 14 days after vaccination as measured by ELISpot assay were reported. RSV F specific T-cell IFN gamma ELISpot responses were measured as counts of spot forming cells per million peripheral blood mononuclear cells (SFC/10^6 PBMCs).
Time Frame: 14 days post vaccination on Day 1 (Day 15)
Population: PPI population included all randomized and vaccinated participants who were part of the immuno subset and for whom immunogenicity data were available. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: SFC/10^6 PBMCs
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 185 | 92
SFC/10^6 PBMCs | 533 [306 to 873] | NA [NA to 78] — Median and lower limit of full range could not be estimated as it was below the lower limit of quantification (LLOQ: 68 SFC/10^6 PBMCs ).

14. Secondary Outcome: Area Under the Curve (AUC) of the Change From Baseline in Respiratory Infection Intensity and Impact Questionnaire (RiiQ) Total Symptom Scale Score
Description: RiiQ symptom scale was a 13-items questionnaire rated on a 4-point scale. The respiratory symptoms included 2 upper respiratory tract infection (URTI) symptoms (nasal congestion and sore throat), 4 lower respiratory tract infection (LRTI) symptoms (cough, wheezing, short of breath, and coughing up phlegm/sputum) and 7 systemic symptoms (headache, feeling feverish, neck pain, body aches and pain, fatigue/tiredness, interrupted sleep, and loss of appetite). Each symptom was rated on a scale of 0 to 3 where 0=None, 1=Mild, 2=Moderate, and 3=Severe. Higher scores indicated greater severity. RiiQ total Symptom score was the mean of all scores (based on 13 symptoms). The AUC of the change from baseline for the RiiQ total symptom score and the RiiQ lower respiratory symptom score during the ARI was calculated.
Time Frame: Baseline (Day 1) up to 24 months
Population: PPE population includes all randomized and vaccinated participants, excluding those with major protocol deviations (MPDs) expecting to impact the efficacy outcomes. Participants with an RSV onset within 14 days after vaccination and participants who discontinued within 14 days after vaccination were excluded from the PPE population. Here, 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Scores on a scale*hours
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
Number analyzed (Participants) | 115 | 143
Scores on a scale*hours | 82 [21 to 141] | 107 [48 to 218]

ADVERSE EVENTS:
Time Frame: From Day 1 up to 24 months post-vaccination on Day 1 (Day 731).
Description: All-cause mortality and serious adverse events (SAEs) were analyzed on Full Analysis Set (FAS) population. Other (not including serious) AEs as solicited and unsolicited AEs were collected and analyzed on a subset of FAS that is called safety subset. The safety subset included all participants that consented to the collection of AEs (solicited and unsolicited AEs).
Arm/Group | Group 1: Ad26.RSV.preF and RSV preF Protein | Group 2: Placebo
All-Cause Mortality (participants affected / at risk) | 105/16709 | 61/8367
Serious Adverse Events (participants affected / at risk) | 842/16709 | 457/8367
Other Adverse Events (participants affected / at risk) | 1477/2330 | 408/1165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.RSV.preF and RSV preF Protein (N=16709) | Group 2: Placebo (N=8367)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 1 (1)
Anaemia Megaloblastic (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenopathy Mediastinal (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Acute Coronary Syndrome (Cardiac disorders) | 1 (1) | 0 (0)
Acute Left Ventricular Failure (Cardiac disorders) | 1 (1) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 17 (17) | 10 (10)
Angina Pectoris (Cardiac disorders) | 6 (6) | 2 (2)
Angina Unstable (Cardiac disorders) | 2 (2) | 4 (4)
Aortic Valve Incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Aortic Valve Stenosis (Cardiac disorders) | 0 (0) | 2 (3)
Arrhythmia (Cardiac disorders) | 2 (2) | 2 (2)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 24 (24) | 13 (13)
Atrial Flutter (Cardiac disorders) | 0 (0) | 2 (2)
Atrial Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Complete (Cardiac disorders) | 1 (1) | 0 (0)
Atrioventricular Block Second Degree (Cardiac disorders) | 3 (3) | 0 (0)
Bradyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 8 (8) | 1 (1)
Cardiac Failure (Cardiac disorders) | 7 (7) | 4 (4)
Cardiac Failure Chronic (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac Failure Congestive (Cardiac disorders) | 15 (16) | 6 (7)
Cardiac Valve Disease (Cardiac disorders) | 1 (1) | 1 (1)
Cardiac Ventricular Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Cardio-Respiratory Arrest (Cardiac disorders) | 3 (3) | 1 (1)
Cardiogenic Shock (Cardiac disorders) | 0 (0) | 2 (2)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Chronic Coronary Syndrome (Cardiac disorders) | 1 (2) | 0 (0)
Conduction Disorder (Cardiac disorders) | 0 (0) | 1 (1)
Congestive Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Cor Pulmonale (Cardiac disorders) | 1 (1) | 0 (0)
Cor Pulmonale Chronic (Cardiac disorders) | 2 (2) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 14 (14) | 11 (12)
Coronary Artery Occlusion (Cardiac disorders) | 1 (1) | 1 (1)
Coronary Artery Thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Hypertensive Heart Disease (Cardiac disorders) | 1 (1) | 0 (0)
Interventricular Septum Rupture (Cardiac disorders) | 1 (1) | 0 (0)
Ischaemic Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Disease (Cardiac disorders) | 1 (1) | 0 (0)
Mitral Valve Incompetence (Cardiac disorders) | 3 (3) | 1 (1)
Mitral Valve Stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 23 (24) | 12 (13)
Myocardial Ischaemia (Cardiac disorders) | 1 (1) | 2 (4)
Pericardial Effusion (Cardiac disorders) | 3 (3) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 3 (3)
Sinus Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Stress Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular Tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 3 (4) | 1 (1)
Hypertrophic Cardiomyopathy (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vitello-Intestinal Duct Remnant (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 3 (3)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Myxoedema (Endocrine disorders) | 1 (1) | 0 (0)
Pituitary Cyst (Endocrine disorders) | 0 (0) | 1 (1)
Angle Closure Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Cataract (Eye disorders) | 2 (2) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Ocular Myasthenia (Eye disorders) | 1 (1) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0)
Vision Blurred (Eye disorders) | 1 (1) | 0 (0)
Abdominal Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 5 (5) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (2)
Colitis (Gastrointestinal disorders) | 3 (3) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 1 (1) | 1 (1)
Duodenal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal Ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastric Ulcer (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastric Ulcer Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric Ulcer Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (2)
Gastritis Erosive (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (3) | 0 (0)
Gastrointestinal Ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hiatus Hernia (Gastrointestinal disorders) | 5 (7) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal Hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Inguinal Hernia Strangulated (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 6 (7) | 1 (1)
Intestinal Perforation (Gastrointestinal disorders) | 2 (2) | 1 (1)
Irritable Bowel Syndrome (Gastrointestinal disorders) | 3 (3) | 0 (0)
Large Intestine Perforation (Gastrointestinal disorders) | 2 (2) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 1 (1)
Mesenteric Panniculitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophageal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Rupture (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal Varices Haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 2 (2) | 2 (2)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small Intestinal Obstruction (Gastrointestinal disorders) | 8 (8) | 1 (1)
Small Intestinal Perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Spigelian Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Tongue Dysplasia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 3 (3) | 2 (2)
Accidental Death (General disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 2 (2)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 3 (3) | 4 (4)
Complication Associated with Device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 18 (18) | 18 (18)
Drowning (General disorders) | 1 (1) | 0 (0)
Drug Withdrawal Syndrome (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Hypothermia (General disorders) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple Organ Dysfunction Syndrome (General disorders) | 2 (2) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 2 (2) | 1 (1)
Pain (General disorders) | 1 (2) | 0 (0)
Prosthetic Cardiac Valve Thrombosis (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Sudden Death (General disorders) | 2 (2) | 2 (2)
Vascular Stent Stenosis (General disorders) | 0 (0) | 1 (2)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1) | 1 (1)
Biliary Tract Disorder (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 8 (8)
Cholecystitis Acute (Hepatobiliary disorders) | 4 (4) | 1 (1)
Cholecystitis Chronic (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 3 (3) | 2 (2)
Hepatic Cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatorenal Syndrome (Hepatobiliary disorders) | 0 (0) | 1 (1)
Amyloidosis (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic Reaction (Immune system disorders) | 0 (0) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal Abscess (Infections and infestations) | 0 (0) | 1 (2)
Abscess (Infections and infestations) | 0 (0) | 1 (1)
Abscess Jaw (Infections and infestations) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 3 (4) | 1 (1)
Anal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Anorectal Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 2 (2) | 2 (2)
Appendicitis Perforated (Infections and infestations) | 1 (1) | 0 (0)
Arthritis Bacterial (Infections and infestations) | 2 (2) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 2 (2)
Bacterial Infection (Infections and infestations) | 1 (1) | 0 (0)
Beta Haemolytic Streptococcal Infection (Infections and infestations) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Bronchitis Viral (Infections and infestations) | 0 (0) | 1 (1)
Carbuncle (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 6 (7) | 5 (5)
Cellulitis Staphylococcal (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Colitis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium Difficile Infection (Infections and infestations) | 1 (1) | 1 (1)
Colonic Abscess (Infections and infestations) | 1 (3) | 2 (2)
Coronavirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Covid-19 (Infections and infestations) | 29 (29) | 12 (12)
Covid-19 Pneumonia (Infections and infestations) | 6 (6) | 4 (4)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Diabetic Foot Infection (Infections and infestations) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 5 (5) | 5 (5)
Diverticulitis Intestinal Perforated (Infections and infestations) | 1 (1) | 0 (0)
Enterococcal Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis Infectious (Infections and infestations) | 1 (1) | 0 (0)
Epiglottic Abscess (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Escherichia Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Extradural Abscess (Infections and infestations) | 0 (0) | 1 (1)
Fungaemia (Infections and infestations) | 1 (1) | 0 (0)
Gangrene (Infections and infestations) | 2 (2) | 0 (0)
Gastroenteritis (Infections and infestations) | 5 (5) | 2 (2)
Gastroenteritis Salmonella (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis Viral (Infections and infestations) | 1 (1) | 0 (0)
Helicobacter Gastritis (Infections and infestations) | 0 (0) | 1 (1)
Herpes Zoster (Infections and infestations) | 3 (3) | 0 (0)
Infected Bite (Infections and infestations) | 1 (1) | 0 (0)
Infected Skin Ulcer (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0)
Infectious Pleural Effusion (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 4 (4)
Intervertebral Discitis (Infections and infestations) | 2 (2) | 0 (0)
Kidney Infection (Infections and infestations) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 1 (1) | 0 (0)
Localised Infection (Infections and infestations) | 3 (3) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 7 (8) | 3 (3)
Lung Abscess (Infections and infestations) | 1 (1) | 1 (1)
Meningoencephalitis Herpetic (Infections and infestations) | 0 (0) | 1 (1)
Metapneumovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 2 (2) | 2 (2)
Perirectal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis Streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 46 (48) | 26 (26)
Pneumonia Aspiration (Infections and infestations) | 5 (5) | 2 (2)
Pneumonia Bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia Influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia Legionella (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia Streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Abscess (Infections and infestations) | 0 (0) | 1 (1)
Postoperative Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0)
Renal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Rhinovirus Infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 15 (15) | 9 (10)
Septic Shock (Infections and infestations) | 4 (4) | 3 (3)
Sinusitis Fungal (Infections and infestations) | 1 (1) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal Sepsis (Infections and infestations) | 1 (1) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 7 (10) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 3 (3)
Viral Labyrinthitis (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol Poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 4 (4)
Arterial Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Asbestosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Bone Contusion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Clavicle Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Craniocerebral Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Extradural Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Eye Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Face Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Facial Bones Fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 5 (5) | 4 (4)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Femur Fracture (Injury, poisoning and procedural complications) | 8 (9) | 5 (5)
Fibula Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Forearm Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Foreign Body in Skin or Subcutaneous Tissue (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Hip Fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Humerus Fracture (Injury, poisoning and procedural complications) | 4 (4) | 3 (3)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint Dislocation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Joint Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament Rupture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Liver Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Meniscus Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
Neck Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Patella Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pelvic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Periprocedural Myocardial Infarction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Periprosthetic Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Pneumothorax Traumatic (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post Vaccination Syndrome (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative Ileus (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural Complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural Pain (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Radius Fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib Fracture (Injury, poisoning and procedural complications) | 10 (10) | 4 (4)
Road Traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Subdural Haematoma (Injury, poisoning and procedural complications) | 6 (7) | 1 (1)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Tendon Rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Tibia Fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Traumatic Haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Haemothorax (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic Intracranial Haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Traumatic Lung Injury (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Body Temperature Increased (Investigations) | 1 (1) | 0 (0)
Cardiac Murmur (Investigations) | 1 (1) | 0 (0)
Computerised Tomogram Thorax Abnormal (Investigations) | 1 (1) | 0 (0)
Electrocardiogram Abnormal (Investigations) | 1 (2) | 0 (0)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1)
Human Metapneumovirus Test Positive (Investigations) | 1 (1) | 0 (0)
Sars-Cov-2 Test Positive (Investigations) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (6) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 4 (4) | 3 (4)
Electrolyte Imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Failure to Thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Lactic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Type 2 Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Cervical Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Inclusion Body Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Degeneration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 16 (16) | 13 (14)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoporotic Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Soft Tissue Necrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Spinal Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Vertebral Foraminal Stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Acute Promyelocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Adenocarcinoma of Colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (3)
Benign Renal Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0)
Bile Duct Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Bladder Squamous Cell Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bowen's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Brain Stem Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 11 (11) | 2 (2)
Breast Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cerebral Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Chronic Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Colon Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 3 (3)
Colon Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Colorectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 0 (0)
Desmoplastic Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Diffuse Large B-Cell Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Endometrial Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial Cancer Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial Cancer Stage Ii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Glioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hepatic Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Hodgkin's Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intestinal Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Intraductal Proliferative Breast Lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3) | 0 (0)
Invasive Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (2)
Invasive Lobular Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Large Intestine Benign Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Laryngeal Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lung Carcinoma Cell Type Unspecified Stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung Carcinoma Cell Type Unspecified Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Lymphocytic Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Malignant Melanoma Stage Iii (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant Melanoma in Situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (4) | 0 (0)
Metastatic Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastatic Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastatic Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Mucinous Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-Hodgkin's Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Small Cell Lung Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oesophageal Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 3 (3)
Pancreatic Carcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Pancreatic Carcinoma Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pituitary Tumour Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Plasma Cell Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Pleomorphic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Polycythaemia Vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Prostate Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 18 (18) | 4 (4)
Prostate Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Rectal Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Rectal Cancer Stage Iv (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Renal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Skin Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Cell Lung Cancer Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small Intestine Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous Cell Carcinoma of Lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Tonsil Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Urethral Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Vaginal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 1 (1)
Balance Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Basal Ganglia Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Bell's Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Brain Injury (Nervous system disorders) | 0 (0) | 1 (1)
Carotid Artery Disease (Nervous system disorders) | 1 (1) | 0 (0)
Carotid Artery Stenosis (Nervous system disorders) | 0 (0) | 1 (2)
Cerebellar Stroke (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 2 (2) | 2 (2)
Cerebral Infarction (Nervous system disorders) | 9 (9) | 3 (3)
Cerebral Mass Effect (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral Venous Sinus Thrombosis (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrospinal Fluid Leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular Accident (Nervous system disorders) | 20 (20) | 8 (8)
Cerebrovascular Disorder (Nervous system disorders) | 1 (1) | 0 (0)
Cervical Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Diabetic Neuropathy (Nervous system disorders) | 3 (3) | 0 (0)
Dizziness Postural (Nervous system disorders) | 1 (1) | 0 (0)
Embolic Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 0 (0) | 2 (2)
Haemorrhagic Stroke (Nervous system disorders) | 2 (2) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Hepatic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Intracranial Aneurysm (Nervous system disorders) | 0 (0) | 2 (3)
Intracranial Mass (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic Stroke (Nervous system disorders) | 7 (7) | 7 (7)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0)
Lacunar Stroke (Nervous system disorders) | 0 (0) | 2 (2)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar Radiculopathy (Nervous system disorders) | 1 (1) | 1 (1)
Lumbosacral Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Monoplegia (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia Gravis (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenic Syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Myelopathy (Nervous system disorders) | 0 (0) | 1 (1)
Nerve Compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 2 (2) | 0 (0)
Ophthalmic Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Parkinson's Disease (Nervous system disorders) | 0 (0) | 1 (1)
Partial Seizures (Nervous system disorders) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Progressive Supranuclear Palsy (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 3 (4)
Spinal Claudication (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid Haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 7 (7) | 7 (7)
Toxic Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Transient Global Amnesia (Nervous system disorders) | 2 (2) | 0 (0)
Transient Ischaemic Attack (Nervous system disorders) | 15 (15) | 11 (11)
Trigeminal Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Vascular Dementia (Nervous system disorders) | 1 (1) | 0 (0)
Vertigo CNS Origin (Nervous system disorders) | 0 (0) | 1 (1)
Device Dislocation (Product Issues) | 1 (1) | 1 (1)
Device Loosening (Product Issues) | 1 (1) | 1 (1)
Device Malfunction (Product Issues) | 0 (0) | 1 (1)
Device Pacing Issue (Product Issues) | 0 (0) | 1 (1)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Confusional State (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 1 (1)
Drug Abuse (Psychiatric disorders) | 1 (1) | 0 (0)
Major Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 1 (1) | 0 (0)
Neurosis (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 2 (2) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 7 (7) | 5 (5)
Chronic Kidney Disease (Renal and urinary disorders) | 2 (2) | 2 (2)
End Stage Renal Disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 2 (2) | 1 (1)
Nephritic Syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 4 (4) | 4 (4)
Prerenal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Failure (Renal and urinary disorders) | 2 (2) | 1 (2)
Renal Haemorrhage (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal Mass (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureterolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral Caruncle (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary Tract Disorder (Renal and urinary disorders) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 3 (3) | 4 (5)
Ovarian Cyst (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Uterine Prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterovaginal Prolapse (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Acute Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 18 (19) | 7 (7)
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6)
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 31 (33) | 14 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cystic Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pharyngeal Mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 5 (5)
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 29 (29) | 9 (9)
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary Thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Sinus Disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3)
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Loss of Personal Independence in Daily Activities (Social circumstances) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 1 (1) | 0 (0)
Aortic Aneurysm (Vascular disorders) | 4 (5) | 1 (1)
Aortic Dissection (Vascular disorders) | 1 (1) | 1 (1)
Aortic Stenosis (Vascular disorders) | 2 (2) | 1 (1)
Arterial Occlusive Disease (Vascular disorders) | 1 (1) | 1 (1)
Arteriosclerosis (Vascular disorders) | 3 (3) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 15 (17) | 3 (3)
Extravasation Blood (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 6 (6) | 0 (0)
Hypertensive Crisis (Vascular disorders) | 1 (1) | 0 (0)
Hypertensive Emergency (Vascular disorders) | 2 (2) | 0 (0)
Hypertensive Urgency (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 5 (5) | 2 (2)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Arterial Occlusive Disease (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Artery Aneurysm (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Artery Stenosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Artery Thrombosis (Vascular disorders) | 2 (2) | 0 (0)
Peripheral Ischaemia (Vascular disorders) | 1 (1) | 0 (0)
Peripheral Vascular Disorder (Vascular disorders) | 1 (1) | 0 (0)
Shock (Vascular disorders) | 1 (1) | 1 (1)
Shock Haemorrhagic (Vascular disorders) | 1 (1) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0)
Venous Thrombosis Limb (Vascular disorders) | 0 (0) | 1 (1)
White Coat Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Ad26.RSV.preF and RSV preF Protein (N=2330) | Group 2: Placebo (N=1165)
Nausea(Solicited) (Gastrointestinal disorders) | 324 (324) | 75 (75)
Fatigue(Solicited) (General disorders) | 789 (789) | 165 (165)
Pain (General disorders) | 48 (61) | 12 (18)
Pyrexia(Solicited) (General disorders) | 171 (171) | 5 (5)
Vaccination Site Erythema(Solicited) (General disorders) | 63 (63) | 5 (5)
Vaccination Site Pain(Solicited) (General disorders) | 1065 (1065) | 168 (168)
Vaccination Site Swelling(Solicited) (General disorders) | 68 (68) | 3 (3)
Blood Pressure Diastolic Increased (Investigations) | 58 (58) | 21 (21)
Blood Pressure Systolic Increased (Investigations) | 150 (150) | 60 (60)
Respiratory Rate Increased (Investigations) | 89 (89) | 49 (49)
Myalgia(Solicited) (Musculoskeletal and connective tissue disorders) | 614 (614) | 119 (119)
Headache(Solicited) (Nervous system disorders) | 597 (597) | 128 (128)
Cough (Respiratory, thoracic and mediastinal disorders) | 68 (74) | 25 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/83/NCT04908683/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-05): https://cdn.clinicaltrials.gov/large-docs/83/NCT04908683/SAP_001.pdf